CLINICAL TRIAL: NCT05782140
Title: ALgorithms Adapted From Remote Monitoring
Acronym: ALARM
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Janani S. Reisenauer, Assistant Professor of Surgery, College of Medicine, Mayo Clinic
Other Study IDs: 22-003308
Record Dates: First submitted 2023-02-24; First posted 2023-03-23 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Surgery
Keywords: Remote Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mayo Clinic Rochester Surgical Patients: Mayo Clinic Watch Device
  Interventions: Device: Mayo Clinic Watch Device

INTERVENTIONS:
Device: Mayo Clinic Watch Device — Mayo Clinic remote monitoring platform (Omni) that utilizes a wearable device with integrated physiological monitoring capabilities.

SUMMARY:
Through the aid of remote monitoring and early symptom detection, a patient's response to stress and normalization to their individual baseline can better contribute towards algorithms which are predictive of clinical decline.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Scheduled to undergo surgery resulting in a complex recovery as evaluated by the treating Department of Surgery surgeon. This includes but is not limited to the following inpatient elective surgery procedures: esophagectomy, pancreatectomy, major liver resections, open vascular surgery, lower extremity bypass, colectomy, and complex pulmonary resections (lobes and above).
* Subjects are committed to daily exercise as outlined in the protocol.

Exclusion Criteria:

* <18 years of age
* Subject is pregnant
* Subject is dismissed from the hospital to a nursing home or long term care facility.
* Subject cannot commitment to daily exercise as outlined in the protocol.
* Subjects enrolled in another device or drug study does not necessarily preclude them from participating in this study. Please check with the PI for inclusion if the subject is on another device or drug study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing surgery in the Mayo Clinic Rochester Department of Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Compliance of Remote Monitoring | Pre-operative to 15 days post discharge.
  Determine the feasibility of remote monitoring for preoperative assessment and postoperative follow up by evaluation of rate of compliance of physiological monitoring data and patinet recorded logs.

SECONDARY OUTCOMES:
Correlation of Compensatory Reserve Algorithm | Pre-operative to 15 days post discharge.
  Evaluation of compensatory reserve algorithm using collected PPG waveforms by passing the collected waveforms of individuals through the algorithm to determine correlation of its performance particularly related to any events that occur during the postoperative and recovery periods.

CONTACTS AND LOCATIONS:
Overall Officials: Janani Reisenauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials